CLINICAL TRIAL: NCT06731556
Title: Intranasal Diclofenac Sodium, Ibuprofen, and Paracetamol for Pain Relief After Pediatric Tonsillectomy
Brief Title: Analgesic Effects of Intranasal Diclofenac Sodium, Ibuprofen, and Paracetamol in Pediatric Tonsillectomy Cases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20.08.2021-E.28962
Record Dates: First submitted 2024-11-26; First posted 2024-12-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Tonsil Disease; Pain Management; Intranasal Drug Administration
Keywords: Intranasal Spray; intranasal Analgesia; Diclofenac Sodium; Ibuprofen; Paracetamol; Tonsillectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: prospective, randomized study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intranasal Paracetamol (Experimental): Participants in this arm received intranasal paracetamol (1.25 mg/mL) for postoperative pain control. Pain levels were assessed using the Modified CHEOPS scale and the Wong-Baker VAS for children aged 4-8 years, and the standard VAS for children aged 9-15 years. Assessments were performed at 15, 30, 60, 120 minutes, and 2, 4, 6, and 12 hours post-surgery.
  Interventions: Drug: Intranasal Paracetamol
- Intranasal Diclofenac Sodium (Experimental): Participants in this arm received intranasal diclofenac sodium (0.0625 mg/mL) for postoperative pain control. Pain levels were assessed using the Modified CHEOPS scale and the Wong-Baker VAS for children aged 4-8 years, and the standard VAS for children aged 9-15 years. Assessments were performed at 15, 30, 60, 120 minutes, and 2, 4, 6, and 12 hours post-surgery.
  Interventions: Drug: Intranasal Diclofenac Sodium
- Intranasal Ibuprofen (Experimental): Participants in this arm received intranasal ibuprofen (0.375 mg/mL) for postoperative pain control. Pain levels were assessed using the Modified CHEOPS scale and the Wong-Baker VAS for children aged 4-8 years, and the standard VAS for children aged 9-15 years. Assessments were performed at 15, 30, 60, 120 minutes, and 2, 4, 6, and 12 hours post-surgery.
  Interventions: Drug: Intranasal Ibuprofen
- Intravenous Paracetamol (Active Comparator): Participants in this arm received intravenous paracetamol (20 mg/kg/day, twice daily) for postoperative pain control. Pain levels were assessed using the Modified CHEOPS scale and the Wong-Baker VAS for children aged 4-8 years, and the standard VAS for children aged 9-15 years. Assessments were performed at 15, 30, 60, 120 minutes, and 2, 4, 6, and 12 hours post-surgery.
  Interventions: Drug: Intravenous paracetamol

INTERVENTIONS:
Drug: Intravenous paracetamol — Paracetamol was administered intravenously at a dose of 20 mg/kg/day, twice daily.
  Other Names: intravenous paracetamol (Group 4)
  Arms: Intravenous Paracetamol
Drug: Intranasal Paracetamol — Paracetamol at a concentration of 1.25 mg/mL was administered intranasally.
  Arms: Intranasal Paracetamol
Drug: Intranasal Diclofenac Sodium — Diclofenac sodium at a concentration of 0.0625 mg/mL was administered intranasally.
  Arms: Intranasal Diclofenac Sodium
Drug: Intranasal Ibuprofen — Ibuprofen at a concentration of 0.375 mg/mL was administered intranasally.
  Arms: Intranasal Ibuprofen

SUMMARY:
This study aims to evaluate the efficacy and safety of intranasal Diclofenac Sodium, intranasal Ibuprofen, and intranasal Paracetamol for pain control following tonsillectomy in pediatric patients.

DETAILED DESCRIPTION:
Postoperative pain management in pediatric tonsillectomy remains a challenge, with concerns about the safety and efficacy of available analgesic options. Intranasal administration of nonsteroidal anti-inflammatory drugs presents a promising alternative for effective pain relief with minimal side effects.

This prospective, randomized study evaluated the efficacy and safety of intranasal diclofenac sodium, intranasal ibuprofen, and intranasal paracetamol compared to intravenous paracetamol in pediatric patients following tonsillectomy. Sixty patients, aged 2 to 14 years, were divided into four groups to receive either intranasal paracetamol (Group 1), intranasal diclofenac sodium (Group 2), intranasal ibuprofen (Group 3), or intravenous paracetamol (Group 4). Pain was assessed using the CHEOPS, VAS, and Wong-Baker modified VAS scoring systems at various postoperative time points. Statistical analysis was performed using the Kruskal-Wallis and Dunn's tests.

ELIGIBILITY:
Inclusion Criteria:

-Pediatric patients who have undergone a tonsillectomy.

Exclusion Criteria:

* Chronic sinusitis
* Common cold or rhinitis
* Turbinate hypertrophy
* Nasal polyposis
* Deviated nasal septum
* Impaired mucociliary clearance
* Atrophic rhinitis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale measurements | Pain levels were assessed at predefined time points (15, 30, 60, 120 minutes, and 2, 4, 6, 12 hours after surgery).
  CHEOPS consists of a total of 6 categories of behaviour, with specific score ranges for each. The total score ranges from 6 to 16. A score of 16 means a lot of pain, while 4 means no pain.

SECONDARY OUTCOMES:
VISUAL ANALOGUE Scale measurements | Pain levels were assessed at predefined time points (15, 30, 60, 120 minutes, and 2, 4, 6, 12 hours after surgery).
  The patient indicates the level of pain by marking it on a visual scale, with one end of the line labelled 'No Pain' (0) and the other end labelled 'Intolerable Pain' (10).
  0: No pain at all. 1-3: Mild pain. 4-6: Moderate pain. 7-10: Severe pain.

OTHER OUTCOMES:
Wong-Baker Facial Pain Scale (Modified VAS) measurements | Pain levels were assessed at predefined time points (15, 30, 60, 120 minutes, and 2, 4, 6, 12 hours after surgery).
  It is an adapted version for children. Pain is graded on the basis of different facial expressions (happy face → crying face). A happy face means no pain, while a crying face means a lot of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramazan Bahadır KÜÇÜK, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I plan to share the excel file where the results are collected and made understandable
Supporting Information: SAP, ICF
Access Criteria: The period of completion of the study and data analysis 30 December 2024-15 January 2025

DOCUMENTS (3):
  • Study Protocol (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT06731556/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT06731556/SAP_001.pdf
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT06731556/ICF_002.pdf